CLINICAL TRIAL: NCT05059431
Title: The Effect of Human Prostate Tissue on Platelet CD40 Ligand, Toll-like Receptor 4, P-selectin and Platelet-Leukocyte Aggregation: an In Vitro Study
Brief Title: The Effect of Human Prostate Tissue on Platelet Activation
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Wei-Hung Chan, Tri-Service General Hospital, Tri-Service General Hospital
Other Study IDs: 2-103-05-041
Record Dates: First submitted 2021-09-19; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Prostate Hyperplasia; Coagulation; Intravascular; Thrombotic Disorder
Keywords: TURP; coagulopathy; DIC; thrombotic disorder
MeSH Terms: conditions — Prostatic Hyperplasia; Thrombosis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Prostate tissue; blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transurethral resection of the prostate (TURP) is a common and standard urological surgical procedure for managing benign prostatic hyperplasia (BPH). Although surgical technology improved in recent decades, severe complications such as TURP syndrome, hematuria, and postoperative hemorrhage were still considerable. Coagulopathy is one of rare but devastating complication which may contribute to bleeding during and after TURP. Although the exact pathophysiological condition of coagulopathy is not clear, there are several possible mechanisms of TURP associated coagulopathy including: urokinase- (u-PA) and tissue-type plasminogen activator (t-PA)-related fibrinolysis; absorption of irrigating fluid associated dilutional coagulopathy; release of prostatic particles rich in tissue thromboplastins into the circulation causing secondary ﬁbrinolysis and disseminated intravascular coagulopathy (DIC); sepsis with DIC associated with bacteria entering the circulation due to prostatic venous sinuses opening and the using of high pressure irrigation. On the other hand, platelet are essential to hemostasis and thrombosis and its activation also contributes to leukocyte recruitment and DIC. Furthermore, previous studies demonstrated that activated platelets could express TLR4, CD40L, P-selectin and induce platelet-leukocyte aggregation (PLA), which were considered important for systemic inflammatory responses and DIC development. Currently, no study investigating the association of prostate particle and platelet activation. Here, we tested the hypothesis that prostate tissue may induce inflammatory responses through platelet activation by measuring the expression of TLR4, CD40L, P-selectin and PLA on platelets.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for TURP surgery

Exclusion Criteria:

* morbid obesity, bedridden, thromboembolic disease, sepsis, nephrotic syndrome, trauma, malignant tumor, disease associated with increasing blood viscosity.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40-80 year old male scheduled for transurethral resection of the prostate surgery.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

PRIMARY OUTCOMES:
TLR4, CD40L and P-selectin expression | 2 hour, during surgical period
  the expression of platelet activation markers by measuring the mean fluorescence intensity of CD40 ligand, Toll-like receptor 4, P-selectin on platelet surface
Platelet leukocyte aggregation | 2 hour, during surgical period
  measuring platelet-leukocyte aggregation by flow cytometry